CLINICAL TRIAL: NCT05618028
Title: A First-in-Human Study of ABBV-525 (MALT1 Inhibitor) in B-Cell Malignancies
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity in Adult Participants With B-Cell Malignancies Receiving Oral ABBV-525 Tablets
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-324; 2022-503136-13 (Other: EU CT)
Record Dates: First submitted 2022-11-14; First posted 2022-11-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; Chronic Lymphocytic Leukemia; B Cell Malignancies; Non-Hodgkin's Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; B-cell Malignancies; Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma; ABBV-525; Cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-525 Dose Escalation (Experimental): Participants will receive escalating doses of ABBV-525 until doses for optimization are determined, as part of an approximately 64 month study period.
  Interventions: Drug: ABBV-525
- ABBV-525 Dose Optimization (Experimental): Participants will receive one of two doses of ABBV-525 until the recommended phase 2 dose (RP2D) is determined, as part of an approximately 64 month study period.
  Interventions: Drug: ABBV-525
- ABBV-525 Dose Expansion (Experimental): Participants will receive the RP2D dose of ABBV-525, as part of an approximately 64 month study period.
  Interventions: Drug: ABBV-525

INTERVENTIONS:
Drug: ABBV-525 — Oral; Tablet

SUMMARY:
B-cell malignancies are a group of cancers of B lymphocytes, a type of white blood cell responsible for fighting infections. The purpose of this study is to assess safety, tolerability, pharmacokinetics and preliminary efficacy of ABBV-525 as a monotherapy.

ABBV-525 is an investigational drug being developed for the treatment of B-Cell Malignancies. Study doctors put the participants in groups called treatment arms. Participants will receive ABBV-525 at different doses. Approximately 150 adult participants will be enrolled in the study across sites worldwide.

In part 1 (dose escalation), participants will receive escalating oral doses of ABBV-525. In part 2 (dose optimization), participants will receive one of two oral doses of ABBV-525, until the recommended phase 2 dose (RP2D) is determined. In part 3 (dose expansion), participants will receive the RP2D oral dose of ABBV-525. The estimated duration of the study is up to 64 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation (Part 1) Only: Participants with a documented diagnosis of one of the following third line or later of treatment (3L)+ mature B-cell malignancies, from the World Health Organization (WHO)-defined histologies as defined in the protocol.
* Dose Optimization (Part 2) Only: Participants with documented diagnosis of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) with histology based on WHO criteria, with measurable disease requiring treatment as defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL).
* Dose Expansion (Part 3) Only: Participants with documented diagnosis of one of the 3L+ mature B-cell malignancies based on WHO criteria listed in the protocol, with measurable disease requiring treatment.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2.
* Participant has a life expectancy >= 12 weeks.
* Adequate hematological and hepatic function as defined in the protocol.
* Must have archival or freshly collected tumor tissue for correlative studies before study enrollment.
* Participants with prior central nervous system (CNS) disease that has been effectively treated may be eligible.
* Participants with resolved coronavirus disease 2019 (COVID-19) infection are eligible.

Exclusion Criteria:

* Known active CNS disease, or primary CNS lymphoma.
* Known bleeding disorders.
* Known history of stroke or intracranial hemorrhage within 12 months prior to first dose of study treatment.
* Uncontrolled active systemic infection, or active cytomegalovirus infection.
* Active and/or chronic hepatitis B or C infection and/or the criteria listed in the protocol.
* Known history of human immunodeficiency virus (HIV).
* Known active COVID-19 infection. Participant must not have signs/symptoms associated with COVID-19 infection or known exposure to a confirmed case of COVID-19 infection during screening. If participant has signs/symptoms suggestive of COVID-19 infection, the participant must have a negative molecular (e.g., polymerase chain reaction) test or 3 negative antigen test results at least 24 hours apart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) | Up to Approximately 64 Months
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is defined as any untoward medical occurrence, whether associated with study drug or not, that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event requiring medical or surgical intervention to prevent serious outcome.
Number of Participants With Dose-Limiting Toxicities (DLT) | Up to Approximately 28 Days
  A DLT is defined as any AE for which a clear alternative cause cannot be established (eg, attributed to the disease under study, another disease, or to a concomitant medication by the study investigators or medical monitor).
Number of Tumor Lysis Syndrome (TLS) | Up to Approximately 64 Months
  TLS is confirmed by evaluation of electrolyte and fluid status and renal status including urine output.
Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters | Up to Approximately 64 Months
  Clinical laboratory parameters included tests of hematology, chemistry, urinalysis and prolactin. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Parameters | Up to Approximately 64 Months
  Vital sign parameters included body temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Electrocardiograms (ECG) | Up to Approximately 64 Months
  A standard 12-lead ECG will be performed. The investigator will assess the results for clinical significance.
Maximum Observed Plasma Concentration (Cmax) of ABBV-525 | Up to 12 Months
  Maximum observed plasma concentration of ABBV-525.
Time to Cmax (Tmax) of ABBV-525 | Up to 12 Months
  Time to Cmax of ABBV-525.
Area Under the Plasma Concentration-Time Curve (AUC) of ABBV-525 | Up to 12 Months
  Area under the plasma concentration-time curve of ABBV-525.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Approximately 64 Months
  ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR)/very good partial response (VGPR)/partial response (PR) in participants receiving at least 1 dose of study drug.
Duration of Response (DOR) | Up to Approximately 64 Months
  DOR is defined for participants achieving CR/VGPR/PR as the time from the initial response per Investigator review to disease progression or death of any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (39):
- United States (13):
  - University of California Los Angeles Medical Center /ID# 246357, Los Angeles, California
  - Yale University School of Medicine /ID# 259081, New Haven, Connecticut
  - Mount Sinai Medical Center-Miami Beach /ID# 248251, Miami Beach, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc /ID# 250113, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center /ID# 259872, Indianapolis, Indiana
  - Tulane Cancer Center Clinic /ID# 249586, New Orleans, Louisiana
  - START Midwest /ID# 252359, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 245459, New York, New York
  - Atrium Health Levine Cancer Institute /ID# 246363, Charlotte, North Carolina
  - University Of Cincinnati Medical Center /ID# 262288, Cincinnati, Ohio
  - University of Texas MD Anderson Cancer Center /ID# 245463, Houston, Texas
  - University of Utah Health Hospital /ID# 259924, Salt Lake City, Utah
  - Northwest Medical Specialties - Tacoma /ID# 260376, Tacoma, Washington
- Australia (4):
  - Liverpool Hospital /ID# 260191, Liverpool, New South Wales
  - Orange Health Service /ID# 260473, Orange, New South Wales
  - Monash Health - Monash Medical Centre /ID# 246366, Clayton, Victoria
  - The Alfred Hospital /ID# 248592, Melbourne, Victoria
- Belgium (2):
  - UZ Gent /ID# 246462, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 246461, Leuven, Vlaams-Brabant
- France (2):
  - CHRU Lille - Hopital Claude Huriez /ID# 252054, Lille, Nord
  - IUCT Oncopole /ID# 259409, Toulouse, Occitanie
- Charite Universitaetsmedizin Berlin Campus Virchow-Klinikum /ID# 252062, Berlin, Germany
- Israel (4):
  - Shamir Medical Center /ID# 257711, Beer Ya'akov, Central District
  - Hadassah Medical Center-Hebrew University /ID# 251441, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 251442, Ramat Gan, Tel Aviv
  - Rabin Medical Center. /ID# 257665, Petah Tikva
- South Korea (3):
  - Seoul National University Hospital /ID# 266340, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 266341, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 266415, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 246537, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 245475, Barcelona
  - Hospital Clinic de Barcelona /ID# 246543, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 246540, Madrid
  - Hospital Universitario 12 de Octubre /ID# 246538, Madrid
- Taiwan (2):
  - China Medical University Hospital /ID# 266414, Taichung
  - National Taiwan University Hospital /ID# 266343, Taipei
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust /ID# 245470, Leeds, West Yorkshire
  - The Royal Marsden NHS Foundation Trust /ID# 250324, London
  - The Christie Hospital /ID# 250325, Manchester

IPD SHARING:
Plan to Share IPD: No